CLINICAL TRIAL: NCT04981431
Title: A Randomized, Placebo-controlled, Single-blind, Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics After Single and Multiple Dose of Elinzanetant in Japanese Healthy Female Adult Participants
Brief Title: A Study to Learn How Safe Elinzanetant is, How it Affects the Body, and How it Moves Into, Through and Out of the Body After Single and Multiple Doses in Japanese Healthy Female Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 21774
Record Dates: First submitted 2021-07-05; First posted 2021-07-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Vasomotor Symptoms as a Sex Hormone-dependent Disorder in Women and Men
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Elinzanetant single dose step 1 (Experimental): Each participant will receive a single oral dose of elinzanetant or placebo.
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo
- Elinzanetant single dose step 2 (Experimental): Each participant will receive a single oral dose of elinzanetant or placebo.
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo
- Elinzanetant single dose step 3 (Experimental): Each participant will receive a single oral dose of elinzanetant or placebo.
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo
- Elinzanetant single dose step 4 (Experimental): Each participant will receive a single oral dose of elinzanetant or placebo.
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo
- Elinzanetant single dose step 6 (Experimental): Each participant will receive a single oral dose of elinzanetant or placebo.
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo
- Elinzanetant multiple dose step 5 (Experimental): Each participant will receive multiple doses of elinzanetant or placebo administered once a day for 7 consecutive days.
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo

INTERVENTIONS:
Drug: Elinzanetant (BAY3427080) — Oral administration
Drug: Placebo — Oral administration

SUMMARY:
Researchers are looking for a new way to treat women who have symptoms that are caused by the sex hormonal changes that happen when a woman's body is going through the menopause. These symptoms include Vasomotor Symptoms (VMS) (hot flashes), and changes in blood pressure. Menopause is when women stop having a menstrual cycle, also called a period. During the period, the ovaries increasingly produce less sex hormones as a result of the natural ageing process and related hormonal adjustments. The decline in hormone production can lead to various symptoms which, in some cases, can have a very adverse effect on a menopausal woman's quality of life.

In this study, researchers want to learn more about a new substance called elinzanetant. Elinzanetant was developed to treat symptoms caused by sex hormonal changes. It works by blocking a group of proteins called neurokinins from sending signals to other parts of the body, which play a role in starting the symptoms.

In this study, the researchers will learn how safe elinzanetant is and how it affects the body of healthy Japanese women compared to a placebo. A placebo is a treatment that looks like a medicine but does not have any medicine in it. Before a new treatment can be given to patients, researchers do studies in healthy participants to learn more about its safety and how it acts in the body.

There will be 2 parts to this study. In Part A, the participants will take a single dose of either elinzanetant or the placebo. In Part B, the participants will take multiple doses of elinzanetant or the placebo. The participants will take each study treatment as capsules by mouth.

The main purpose of this study is to learn how safe elinzanetant is and how it affects the body. To answer this question, the researchers will collect the medical problems the participants have after receiving the treatment and that may or may not be related to the study treatment. These medical problems are also known as "adverse events".

During Part A, the participants will stay at their study site for a total of 9 days. They will take either elinzanetant or the placebo only on Day 1 of their stay. During Part B, the participants will stay at their study site for a total of 15 days. They will take either elinzanetant or the placebo once a day for 7 days of their stay. Each participant will be in the study for a total of approximately 5 weeks for Part A and approximately 6 weeks for Part B.

During the study, the doctors will:

* take blood and urine samples;
* check the participants' health;
* ask the participants questions about what medicines they are taking and if they are having adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Japanese participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, blood pressure, pulse rate, 12 lead electrocardiogram (ECG), body temperature, and laboratory tests.
* Non-smoker, at least from 3 months before the screening visit onwards.
* Body weight of at least 40 kg and body mass index (BMI) within the range 18.0 and 30.0 kg/m^2 (inclusive).

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Any clinically relevant abnormal findings in medical history and physical examination.
* History or evidence of any clinically relevant cardiovascular, gastrointestinal, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other clinically relevant disease.
* Relevant diseases or febrile illness within the last 4 weeks prior to the first study intervention administration.
* Regular use of medicines, or dietary supplements or other substances, e.g., carnitine products, anabolics, high dose vitamins.
* Use of any systemic or topical medicine or substance within 4 weeks before first study drug intervention, which oppose the study objectives, or which might influence them. This includes medicines and natural remedies (e.g St. John's wort) that are altering the activity of CYP3A4 enzyme and the transporters Breast Cancer Resistance Protein (BCRP) and P-gp.
* ECG: PR interval > 210 msec, QT interval corrected using Bazett's formula (QTcB) >450 msec, QRS duration > 110 msec at screening visit.
* Systolic blood pressure below 90 or above 140 mmHg; diastolic blood pressure below 40 or above 90 mmHg at screening visit.
* Pulse rate below 50 or above 90 beats per minute (bpm; a lower pulse rate between 45 and 50 bpm is acceptable in case of normal thyroid function and absence of symptoms of bradycardia) at screening visit.
* Participants with a presence of any of the following, confirmed by a repeat test: aspartate aminotransferase (AST), alanine aminotransferase (ALT) and/or bilirubin above 1.2 x upper limit of normal (ULN) at screening visit.
* Participants with a presence of gamma-glutamyl transferase (GGT) > ULN confirmed by a repeat test, CK (creatine kinase)>2x ULN, and thyroid-stimulating hormone (TSH) outside normal range at screening visit.
* History of COVID-19 (coronavirus disease 2019).
* Suspected or confirmed active or prior SARS-CoV-2 (severe acute respiratory syndrome coronavirus type 2) infection according to local guidelines/practice.
* Contact with SARS-CoV-2- positive or COVID-19 patient within the last 4 weeks prior to admission to the study site.
* Positive SARS-CoV-2 viral RNA (ribonucleic acid) test.
* Vaccination against SARS-CoV-2 within 14 days before first administration of the study intervention or vaccination planned before completion of the last study visit.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-03-13 (Actual); Study Completion 2022-03-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with and severity of treatment-emergent adverse events (TEAEs) | Up to 2 weeks after start of dosing

SECONDARY OUTCOMES:
Cmax (maximum observed drug concentration after single dose administration) of elinzanetant | Day 1 pre-dose until 144 hours post-dose
  Only for single dose steps 1 to 4 and 6
Cmax/D (Cmax divided by dose) of elinzanetant | Day 1 pre-dose until 144 hours post-dose
  Only for single dose steps 1 to 4 and 6
AUC (area under the concentration vs. time curve from zero to infinity after single dose) of elinzanetant | Day 1 pre-dose until 144 hours post-dose
  Only for single dose steps 1 to 4 and 6
AUC/D (AUC divided by dose) of elinzanetant | Day 1 pre-dose until 144 hours post-dose
  Only for single dose steps 1 to 4 and 6
Cmax,md (maximum observed drug concentration after multiple dose administration) of elinzanetant | Day 7 (pre-dose until 144 hours post-dose)
  Only for multiple dose step 5
Cmax,md/D (Cmax,md divided by dose) of elinzanetant | Day 7 (pre-dose until 144 hours post-dose)
  Only for multiple dose step 5
AUC(0-24)md (AUC from time 0 to 24 h after multiple dose) of elinzanetant | Day 7 (pre-dose until 24 hours post-dose)
  Only for multiple dose step 5
AUC(0-24)md/D (AUC(0-24)md divided by dose) of elinzanetant | Day 7 (pre-dose until 24 hours post-dose)
  Only for multiple dose step 5

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Fukuoka Mirai Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.